CLINICAL TRIAL: NCT06403605
Title: A Randomized Controlled Clinical Trial Evaluating the Efficacy of a Borate-based Bioactive Glass Advanced Wound Matrix and Standard of Care Versus Standard of Care Alone
Brief Title: Bioresorbable Glass Fiber Matrix in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETS Wound Care, LLC (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETS-MG-DFU-02
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer; Ulcer Foot; Diabetic Foot
Keywords: DFU; Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SOC primary dressing with MIRRAGEN™ (Experimental): Mirragen Advanced Wound Matrix is intended for the use in the management of wounds including diabetic ulcers. Wound matrix to be used per manufacturer instructions for use in conjunction with offloading and additional (outer) dressing application with moisture retention dressing.
  Interventions: Device: Mirragen Advanced Wound Matrix
- SOC primary dressing with FIBRACOL™ (Active Comparator): A commercially available wound dressing to be used per manufacturer's instructions for use in conjunction with offloading and additional (outer) dressing application with moisture retention dressing.
  Interventions: Device: Fibracol

INTERVENTIONS:
Device: Mirragen Advanced Wound Matrix — Offloading - patient will be offloaded in a diabetic CAM boot after treatment, or total contact cast if patient cannot be fit in a diabetic boot. Other names; pressure relief.
  Additional "outer" dressing application - application of outer moisture retentive dressing, and a multilayer compression dressing. Other names; outer protective dressing.
  Mirragen Advanced Wound Matrix - application of Mirragen to wound site along with standard of care treatment.
  Arms: SOC primary dressing with MIRRAGEN™
Device: Fibracol — Offloading - patient will be offloaded in a diabetic CAM boot after treatment, or total contact cast if patient cannot be fit in a diabetic boot. Other names; pressure relief.
  Additional "outer" dressing application - application of outer moisture retentive dressing, and a multilayer compression dressing. Other names; outer protective dressing.
  Fibracol - application of Fibracol to wound site along with standard of care treatment.
  Arms: SOC primary dressing with FIBRACOL™

SUMMARY:
This study is a prospective, multi-center, randomized controlled trial designed to collect patient outcome data on 2 commercially available treatments for diabetic foot wounds.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, RCT designed to collect patient outcome data on two commercially available treatments for DFUs. The trial will be single blinded in regard to wound healing assessment (another clinician, other than the investigator at each site will assess wound healing) and confirmation of wound healing will be overseen by an independent adjudication committee made up of wound care experts. The study will last twelve weeks, with a two week screening period prior to enrollment.

There are two arms in the study:

Arm 1: SOC therapy (offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement)) and wound care covering with resorbable bioactive glass fiber, MIRRAGEN™ Advanced Wound Matrix, followed by a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

ARM 2: SOC therapy (offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement)) and wound care covering with calcium alginate Fibracol dressing follwed by a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target diabetic foot ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement with a photographic planimetry app.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be full thickness on the foot or ankle that does not probe to bone.
7. Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

   1. TCOM ≥30 mmHg
   2. ABI between 0.7 and 1.3
   3. PVR: Biphasic
   4. TBI ˃0.6
   5. As an alternative arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to randomization.
10. The subject must consent to using the prescribed off-loading method for the duration of the study.
11. The subject must agree to attend the weekly study visits required by the protocol.
12. The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. A subject known to have a life expectancy of < 6 months is excluded.
2. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
3. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
4. A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
5. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
6. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
7. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
8. If a subject has a glycated hemoglobin (HbA1c) greater than or equal to 12% taken at or within 3 months of the initial screening visit he/she is excluded.
9. If a subject has a serum creatinine ≥ 3.0mg/dL within 6 months of randomization he/she is excluded.
10. The subject is excluded if the surface area measurement of the target ulcer has reduced in size by more than 30% in the 2 weeks prior to the initial screening during the 2-week screening phase: the 2 weeks from the initial screening visit (SV1) to the TV1/randomization visit during which time the subject received SOC.
11. A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
12. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
13. A potential subject with end stage renal disease requiring dialysis is excluded.
14. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days is excluded.
15. A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
16. A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD, PhD, Study Chair — USC/Salsa; Charles M Zelen, DPM, Principal Investigator — Professional Education and Research Institute; Robert Galiano, MD, Study Chair — Professor of Surgery, Plastic Surgery, Northwestern University School of Medicine, Chicago, IL
Locations (15):
- United States (15):
  - LA Foot and Ankle, Los Angeles, California
  - Casa Colina, Pomona, California
  - Center for Clincal Research, San Francisco, California
  - Southernmost Foot and Ankle Specialists, Homestead, Florida
  - Doctor's Research Network, South Miami, Florida
  - Gateway Clinical Trials, O'Fallon, Illinois
  - Foot and Ankle Center of Illinois, Springfield, Illinois
  - Mercy Medical Center, Cedar Rapids, Iowa
  - Foot and Ankle Specialists of the Mid Atlantic, Frederick, Maryland
  - Wound Care Experts, Las Vegas, Nevada
  - Lower Extremity Institute for Research and Therapy, Youngstown, Ohio
  - Wound Centrics, Corpus Christi, Texas
  - PULSE: Amputation Prevention Center, LLC, El Paso, Texas
  - Foot and Ankle Specialists of the Mid Atlantic, Salem, Virginia
  - United Wound Healing P.S, Auburn, Washington

REFERENCES:
- [Result] Armstrong DG, Orgill DP, Galiano RD, Lantis J, Glat PM, Gitterle M, Carter MJ, Young N, Zelen CM. A Borate-Based Bioactive Glass Advances Wound Healing in Non-Healing Wagner Grade 1 Diabetic Foot Ulcers: A Randomised Controlled Clinical Trial. Int Wound J. 2025 Oct;22(10):e70763. doi: 10.1111/iwj.70763. PMID 41014175

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 245 subjects were assessed for eligibility to participate in the study.
Period: Randomization and Initial Treatment
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Started | 77 | 71
Completed | 77 | 71
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Started | 77 | 71
Completed | 52 | 43
Not Completed | 25 | 28
Not completed — Withdrawn per protocol with PAR <50% at week 6 | 17 | 19
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Other reasons | 0 | 4

BASELINE CHARACTERISTICS:
Population: Both modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC Primary Dressing With MIRRAGEN™ | SOC Primary Dressing With FIBRACOL™ | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Both mITT and PP shown.
  years
    mITT | 60.1 (16.81) | 59.1 (14.26) | 59.6 (15.50)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 60.2 (16.34) | 57.7 (15.60) | 59.1 (15.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: Female | 20 | 18 | 38
    mITT: Male | 47 | 48 | 95
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Female | 11 | 9 | 20
    PP: Male | 33 | 29 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: American Indian or Alaska Native | 0 | 0 | 0
    mITT: Asian | 1 | 0 | 1
    mITT: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    mITT: Black or African American | 7 | 4 | 11
    mITT: White | 57 | 60 | 117
    mITT: More than one race | 0 | 0 | 0
    mITT: Unknown or Not Reported | 2 | 2 | 4
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: American Indian or Alaska Native | 0 | 0 | 0
    PP: Asian | 1 | 0 | 1
    PP: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    PP: Black or African American | 5 | 2 | 7
    PP: White | 37 | 34 | 71
    PP: More than one race | 0 | 0 | 0
    PP: Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: Hispanic or Latino | 19 | 14 | 33
    mITT: Not Hispanic or Latino | 48 | 52 | 100
    mITT: Unknown or Not Reported | 0 | 0 | 0
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Hispanic or Latino | 10 | 9 | 19
    PP: Not Hispanic or Latino | 34 | 29 | 63
    PP: Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m²] — Population: Both mITT and PP shown.
  kg/m²
    mITT | 33.9 (8.45) | 35.0 (8.98) | 34.5 (8.71)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 34.3 (9.06) | 36.4 (9.99) | 35.3 (9.50)
Tobacco use [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: Current | 13 | 8 | 21
    mITT: Former | 20 | 22 | 42
    mITT: Never used tobacco | 34 | 36 | 70
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Current | 8 | 4 | 12
    PP: Former | 13 | 15 | 28
    PP: Never used tobacco | 23 | 19 | 42
Diabetes duration [Mean (Standard Deviation); unit: years] — Population: Both mITT and PP shown.
  years
    mITT | 17.1 (13.59) | 15.9 (9.58) | 16.5 (11.71)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 15.7 (9.75) | 16.4 (14.18) | 16.0 (11.93)
Age when first DFU appeared [Mean (Standard Deviation); unit: years] — Population: Both mITT and PP shown.
  years
    mITT | 58.2 (11.56) | 53.6 (11.60) | 55.9 (11.76)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 58.9 (11.86) | 54.4 (11.09) | 56.8 (11.66)
Number of prior DFUs [Mean (Standard Deviation); unit: DFUs] — Population: Both mITT and PP shown.
  DFUs
    mITT | 3.1 (4.27) | 4.4 (4.96) | 3.8 (4.66)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 2.5 (2.95) | 3.6 (3.77) | 3.0 (3.38)
Number of other concurrent DFUs at screening [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: 0 | 48 | 53 | 101
    mITT: 1 | 1 | 0 | 1
    mITT: 2 | 15 | 9 | 24
    mITT: 3 or more | 3 | 4 | 7
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: 0 | 32 | 29 | 61
    PP: 1 | 0 | 0 | 0
    PP: 2 | 11 | 7 | 18
    PP: 3 or more | 1 | 2 | 3
History of DFU recurrence [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 32 | 31 | 63
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 18 | 16 | 34
Major amputation [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 2 | 5 | 7
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 1 | 4 | 5
Minor amputations [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: 0 | 41 | 37 | 78
    mITT: 1 | 11 | 14 | 25
    mITT: 2 | 5 | 7 | 12
    mITT: 3 or more | 10 | 8 | 18
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: 0 | 31 | 21 | 52
    PP: 1 | 6 | 10 | 16
    PP: 2 | 3 | 3 | 6
    PP: 3 or more | 4 | 4 | 8
Major foot deformities [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: Charcot | 5 | 8 | 13
    mITT: Hammertoe | 2 | 1 | 3
    mITT: Varus ankle | 1 | 0 | 1
    mITT: Hallux valgis | 2 | 1 | 3
    mITT: Cavus foot | 3 | 1 | 4
    mITT: None of the above | 54 | 55 | 109
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Charcot | 1 | 4 | 5
    PP: Hammertoe | 1 | 1 | 2
    PP: Varus ankle | 0 | 0 | 0
    PP: Hallux valgis | 2 | 1 | 3
    PP: Cavus foot | 2 | 1 | 3
    PP: None of the above | 38 | 31 | 69
Creatinine [Mean (Standard Deviation); unit: mg/dL] — Population: Both mITT and PP shown.
  mg/dL
    mITT | 1.09 (0.42) | 1.24 (0.54) | 1.2 (0.49)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 1.09 (0.46) | 1.19 (0.46) | 1.1 (0.46)
HbA1c [Mean (Standard Deviation); unit: %] — Population: Both mITT and PP shown.
  %
    mITT | 7.7 (1.69) | 7.4 (1.65) | 7.6 (1.67)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 7.7 (1.61) | 7.4 (1.57) | 7.6 (1.60)
Wound area [Mean (Standard Deviation); unit: cm^2] — Population: Both mITT and PP shown.
  cm^2
    mITT | 3.1 (2.81) | 3.3 (2.57) | 3.2 (2.69)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 2.7 (2.37) | 3.1 (2.43) | 2.9 (2.39)
Wound age [Mean (Standard Deviation); unit: weeks] — Population: Both mITT and PP shown.
  weeks
    mITT | 20.9 (13.26) | 20.9 (14.82) | 20.9 (14.00)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 19.4 (12.99) | 21.3 (14.55) | 20.3 (13.69)
Number of participants with index wound in each vertical location [Count of Participants; unit: Participants] — Index ulcer location is defined by the ulcer being on the left or right foot, by the vertical location of the ulcer on the foot (dorsal or plantar), anatomical location (toe, forefoot, midfoot, hind foot, ankle, or heel), and the positioning of the ulcer as lateral or medial located. Population: Both mITT and PP shown.
  Participants
    mITT: Plantar | 52 | 54 | 106
    mITT: Dorsal | 15 | 12 | 27
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Plantar | 34 | 29 | 63
    PP: Dorsal | 10 | 9 | 19
Number of participants with index wound in each position [Count of Participants; unit: Participants] — Index ulcer location is defined by the ulcer being on the left or right foot, by the vertical location of the ulcer on the foot (dorsal or plantar), anatomical location (toe, forefoot, midfoot, hind foot, ankle, or heel), and the positioning of the ulcer as lateral or medial located. Population: Both mITT and PP shown.
  Participants
    mITT: Medial | 35 | 37 | 72
    mITT: Lateral | 32 | 28 | 60
    mITT: Unknown | 0 | 1 | 1
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Medial | 26 | 20 | 46
    PP: Lateral | 18 | 17 | 35
    PP: Unknown | 0 | 1 | 1
Number of participants with index wound in each anatomical location [Count of Participants; unit: Participants] — Index ulcer location is defined by the ulcer being on the left or right foot, by the vertical location of the ulcer on the foot (dorsal or plantar), anatomical location (toe, forefoot, midfoot, hind foot, ankle, or heel), and the positioning of the ulcer as lateral or medial located. Population: Both mITT and PP shown.
  Participants
    mITT: Toe | 13 | 10 | 23
    mITT: Forefoot | 29 | 24 | 53
    mITT: Midfoot | 12 | 17 | 29
    mITT: Hindfoot | 2 | 2 | 4
    mITT: Heel | 9 | 10 | 19
    mITT: Ankle | 2 | 3 | 5
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Toe | 13 | 6 | 19
    PP: Forefoot | 18 | 15 | 33
    PP: Midfoot | 5 | 7 | 12
    PP: Hindfoot | 1 | 1 | 2
    PP: Heel | 6 | 6 | 12
    PP: Ankle | 1 | 3 | 4
Off-loading type [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT: Boot | 10 | 11 | 21
    mITT: CAM boot | 28 | 31 | 59
    mITT: Shoe | 10 | 9 | 19
    mITT: Other | 5 | 2 | 7
    mITT: No off-loading | 14 | 13 | 27
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP: Boot | 6 | 10 | 16
    PP: CAM boot | 21 | 14 | 35
    PP: Shoe | 4 | 3 | 7
    PP: Other | 3 | 2 | 5
    PP: No off-loading | 10 | 9 | 19
Number of debridements [Mean (Standard Deviation); unit: debridements] — Population: Both mITT and PP shown.
  debridements
    mITT | 9.0 (3.54) | 9.2 (3.34) | 9.1 (3.43)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 9.4 (4.09) | 9.7 (3.85) | 9.6 (3.96)
Number of comorbidities [Mean (Standard Deviation); unit: comorbidities] — All identified comorbidities from medical history. Population: Both mITT and PP shown.
  comorbidities
    mITT | 7.1 (5.48) | 7.9 (4.29) | 7.5 (4.92)
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 6.3 (4.50) | 8.0 (4.32) | 7.1 (4.47)
Comorbidities: chronic kidney disease (CKD) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 4 | 11 | 15
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 3 | 5 | 8
Comorbidities: hypertension [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 41 | 49 | 90
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 25 | 25 | 50
Comorbidities: peripheral arterial disease (PAD) / peripheral vascular disease (PVD) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 7 | 5 | 12
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 5 | 5 | 10
Comorbidities: chronic heart failure (CHF) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 4 | 3 | 7
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 4 | 2 | 6
Comorbidities: hyperlipidemia / dyslipidemia [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 20 | 24 | 44
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 14 | 11 | 25
Comorbidities: gastroesophageal reflux disease (GERD) [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 13 | 17 | 30
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 11 | 7 | 18
Comorbidities: hypothyroidism [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 9 | 11 | 20
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 7 | 6 | 13
Comorbidities: lower extremity edema [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 4 | 6 | 10
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 4 | 1 | 5
Comorbidities: peripheral neuropathy [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 27 | 34 | 61
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 19 | 17 | 36
Comorbidities: any psychiatric condition [Count of Participants; unit: Participants] — Population: Both mITT and PP shown.
  Participants
    mITT | 17 | 22 | 39
    PP: number analyzed (Participants) | 44 | 38 | 82
    PP | 13 | 13 | 26

OUTCOME MEASURES:

1. Secondary Outcome: Percentage Area Reduction (PAR)
Description: Percentage wound area reduction measured weekly with digital photographic planimetry and physical examination
Time Frame: 12 weeks
Population: Both the modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Number analyzed (Participants) | 67 | 66
percent
  mITT | 48.8 (82.81) | 53.7 (65.78)
  PP: number analyzed (Participants) | 44 | 38
  PP | 93.7 (15.28) | 89.7 (25.19)
Statistical Analysis 1: Comparison: SOC primary dressing with MIRRAGEN™ vs SOC primary dressing with FIBRACOL™; Test type: Superiority; p = 0.78, Mixed Models Analysis — Adjusted p value in the mITT analysis population
Statistical Analysis 2: Comparison: SOC primary dressing with MIRRAGEN™ vs SOC primary dressing with FIBRACOL™; Test type: Superiority; p = 0.48, Mixed Models Analysis — Adjusted p value in the PP analysis population

2. Secondary Outcome: Time to Heal
Description: The time to achieve complete wound closure within 12 weeks.
Time Frame: 12 weeks
Population: Both the modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Number analyzed (Participants) | 67 | 66
days
  mITT | 63.4 [56.6 to 70.1] | 72.5 [67.3 to 77.7]
  PP: number analyzed (Participants) | 44 | 38
  PP | 57.5 [49.3 to 65.7] | 67.8 [60.5 to 75.2]
Statistical Analysis 1: Comparison: SOC primary dressing with MIRRAGEN™ vs SOC primary dressing with FIBRACOL™; Test type: Superiority; p = 0.049, Log Rank — Adjusted p-value in the mITT population
Statistical Analysis 2: Comparison: SOC primary dressing with MIRRAGEN™ vs SOC primary dressing with FIBRACOL™; Test type: Superiority; p = 0.084, Log Rank — Adjusted p value in the PP population

3. Secondary Outcome: Changes in Quality of Life
Description: The WOUND-Q is a questionnaire measuring outcomes important to patients with chronic wounds. Five of the tool's 13 independently functioning scales (with 5 to 11 items each) were measured in this study. 'Assessment' measures how concerned someone has been with their wound(s). 'Drainage' measures how bothered someone has been by drainage from their wound(s). 'Smell' measures how bothered someone has been by the smell from their wound(s). 'Social' measures the impact of a person's wound(s) on their social life. 'Dressing' measures someone's satisfaction with their wound dressing. For all of these scales, possible responses to each item range from minimum 0 ('not at all') to maximum 4 ('very much'). To score a scale, the raw scores for the set of items in a scale are added together to produce a total raw score. The total raw score for the scale is then converted to a score that ranges from 0 to 100. For all, higher scores represent better outcomes.
Time Frame: 12 weeks
Population: Both the modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Number analyzed (Participants) | 67 | 66
units on a scale
  Assessment (mITT) | 18.3 (20.68) | 17.0 (21.36)
  Drainage (mITT) | 16.6 (22.77) | 11.8 (20.83)
  Smell (mITT) | 4.5 (23.06) | 1.4 (18.42)
  Social (mITT) | 11.6 (28.14) | 15.2 (26.27)
  Dressing (mITT) | 9.0 (21.08) | 7.1 (18.04)
  Assessment (PP): number analyzed (Participants) | 44 | 38
  Assessment (PP) | 28.1 (17.89) | 24.6 (21.34)
  Drainage (PP): number analyzed (Participants) | 44 | 38
  Drainage (PP) | 25.3 (19.58) | 17.6 (18.57)
  Smell (PP): number analyzed (Participants) | 44 | 38
  Smell (PP) | 8.1 (20.73) | 3.4 (17.59)
  Social (PP): number analyzed (Participants) | 44 | 38
  Social (PP) | 17.4 (29.39) | 19.0 (25.53)
  Dressing (PP): number analyzed (Participants) | 44 | 38
  Dressing (PP) | 14.2 (20.85) | 7.7 (18.55)

4. Secondary Outcome: Change in Pain Level
Description: The FACES pain scale was administered to the clinical trial participants at each visit. The trial participant selected their pain level with a series of faces that correspond to a number between 0 which implies no pain, up to 10 which implies the most severe pain.
Time Frame: 12 weeks
Population: Both the modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Measure: Mean (Standard Deviation); unit: score change [EOS - baseline]
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Number analyzed (Participants) | 67 | 66
score change [EOS - baseline]
  mITT | 0.5 (2.47) | 0.8 (2.27)
  PP: number analyzed (Participants) | 44 | 38
  PP | 0.9 (2.24) | 1.0 (2.44)

5. Primary Outcome: Complete Wound Healing
Description: The proportion of subjects achieving complete wound closure.
Time Frame: 12 weeks
Population: Both the modified intent-to-treat (mITT) and per protocol (PP) analysis populations are represented.
Measure: Count of Participants; unit: Participants
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
Number analyzed (Participants) | 67 | 66
Participants
  mITT | 32 | 16
  PP: number analyzed (Participants) | 44 | 38
  PP | 32 | 16
Statistical Analysis 1: Comparison: SOC primary dressing with MIRRAGEN™ vs SOC primary dressing with FIBRACOL™; Test type: Superiority; p = 0.007, Fisher Exact

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up (up to 12 weeks)
Arm/Group | SOC primary dressing with MIRRAGEN™ | SOC primary dressing with FIBRACOL™
All-Cause Mortality (participants affected / at risk) | 1/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 6/67 | 3/66
Other Adverse Events (participants affected / at risk) | 5/67 | 5/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC primary dressing with MIRRAGEN™ (N=67) | SOC primary dressing with FIBRACOL™ (N=66)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) — Not related to receiving the intervention
Deep space infection of left plantar mid foot (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention
Osteomyelitis of sacrum (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention
Postoperative infection of non-study wound (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Necrotizing fasciitis (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Non-study diabetic foot wound infection with osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Death (due to underlying comorbidities) (General disorders) | 1 (1) | 0 (0) — Not related to receiving the intervention
Septicemia (gram negative, from right foot abscess/cellulitis) (Infections and infestations) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Acute toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) — Not related to receiving the intervention.
Cellulitis, right leg (Infections and infestations) | 0 (0) | 1 (1) — Not related to receiving the intervention
Anasarca (Cardiac disorders) | 0 (0) | 1 (1) — Not related to receiving the intervention.
Bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related to receiving the intervention
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related to receiving the intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC primary dressing with MIRRAGEN™ (N=67) | SOC primary dressing with FIBRACOL™ (N=66)
Index wound infection (Infections and infestations) | 5 (5) | 5 (5) — Not including cellulitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT06403605/Prot_SAP_000.pdf